CLINICAL TRIAL: NCT06082531
Title: Therapeutic Effect of Platelet-rich Plasma (PRP) Injection on Knee Osteoarthritis and Periarticular Tissue Injury
Brief Title: Effect of Platelet-rich Plasma (PRP) Injection on Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20232210
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-09

CONDITIONS: Platelets-rich Plasma; Osteoarthritis Knees Both; Meniscus Disorder; Cartilage Injury
Keywords: platelets-rich plasma; Osteoarthritis; Cartilage Injury; Meniscus Injury
MeSH Terms: conditions — Osteoarthritis | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Preoperative (No Intervention)
- postoperative (6 weeks) (Experimental): The patients were injected with PRP.
  Interventions: Drug: Sodium hyaluronate injection
- postoperative (3 months) (Experimental): The patients were injected with PRP.
  Interventions: Drug: Sodium hyaluronate injection

INTERVENTIONS:
Drug: Sodium hyaluronate injection — The control group was injected into the joint cavity with sodium hyaluronate injection..
  Arms: postoperative (3 months); postoperative (6 weeks)

SUMMARY:
To evaluate the safety and effectiveness of PRP injection therapy in the repair of osteoarthritis and periarticular soft tissue injury through a single-center, exploratory clinical study, and to provide a more reliable basis for the treatment of joint injury.

ELIGIBILITY:
Inclusion Criteria:

* The age range of the participants was 20 to 60 years old. Through a comprehensive clinical and imaging examination, it was conclusively determined that the individuals had knee osteoarthritis or experienced injuries to the cart, and meniscus surrounding the knee joint.
* The preoperative routine tests and examinations revealed no contraindications.
* Revised sentence: "Informed consent of the patient

Exclusion Criteria:

* The platelet count or function exhibits significant abnormalities、Systemic infection transmitted through the bloodstream.
* Prolonged usage of anti-inflammatory drugs and systemic corticoid administration.
* In injection site or damage to the skin.
* Patients with tumors or undergoing radiotherapy and chemotherapy.
* Pregnant or breastfeeding women.
* Individuals with mental illnesses who are unable to cooperate with follow-up procedures.
* Contraindications for MRI、Patients or their families do consent to participate in the study.
* Other circumstances that render participation in the study unsuitable.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
X-ray | pre-operation,3 weeks after treatment, 6 months after treatment
  The postoperative plain X-ray film was utilized for the assessment of knee joint deformity, stenosis of the joint space, and hyperplasia of osteophytes.
CT | pre-operation,3 weeks after treatment, 6 months after treatment
  The application of three-dimensional CT scan for the assessment of articular cartilage defects.
MRI | pre-operation,3 weeks after treatment, 6 months after treatment
  The injury of ligaments, meniscus, and the knee joint was assessed using MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramos-Gonzalez G, Salazar L, Wittig O, Diaz-Solano D, Cardier JE. The effects of mesenchymal stromal cells and platelet-rich plasma treatments on cutaneous wound healing. Arch Dermatol Res. 2023 May;315(4):815-823. doi: 10.1007/s00403-022-02451-y. Epub 2022 Nov 3. PMID 36326886
- [Background] Zhang Y, Xing F, Luo R, Duan X. Platelet-Rich Plasma for Bone Fracture Treatment: A Systematic Review of Current Evidence in Preclinical and Clinical Studies. Front Med (Lausanne). 2021 Aug 3;8:676033. doi: 10.3389/fmed.2021.676033. eCollection 2021. PMID 34414200